CLINICAL TRIAL: NCT01193101
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging Study to Evaluate the Efficacy and Safety of LCZ696 Compared to Placebo After 8 Weeks Treatment in Patients With Essential Hypertension
Brief Title: Efficacy and Safety of LCZ696 Compared to Placebo in Patients With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696A2219
Record Dates: First submitted 2010-08-26; First posted 2010-09-01 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure; LCZ696; dual-acting; neprilysin; nep inhibitor; vasopeptidase; angiotensin receptor; ARNi; Essential hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- LCZ696 100 mg (Experimental): LCZ696 100 mg plus placebo daily during double blind (DB) treatment for 8 weeks and then single-blind placebo for one week.
  Interventions: Drug: LCZ696; Drug: Placebo
- LCZ696 200 mg (Experimental): LCZ696 200 mg plus placebo daily during double blind (DB) treatment for 8 weeks and then single-blind placebo for one week.
  Interventions: Drug: LCZ696; Drug: Placebo
- LCZ696 400 mg (Experimental): LCZ696 200 mg LCZ696 plus placebo for one week, then titrated up to 400 mg plus placebo for the remaining 7 weeks during DB treatment, and then single-blind placebo for one week.
  Interventions: Drug: LCZ696; Drug: Placebo
- Placebo (Placebo Comparator): Placebo daily for 8 weeks during DB treatment, and then single-blind placebo for 1 week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LCZ696 — LCZ696
  Arms: LCZ696 100 mg; LCZ696 200 mg; LCZ696 400 mg
Drug: Placebo — matching placebo to LCZ696

SUMMARY:
This study is a phase 2 study in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give written informed consent before any assessment is performed.
2. Patients with mild to moderate essential hypertension, untreated or currently taking antihypertensive therapy (mean sitting diastolic blood pressure ≥ 95 mmHg and < 110 mmHg, and mean sitting systolic blood pressure ≥ 140 mmHg and < 180 mmHg).
3. Patients must be willing and able to undergo ambulatory blood pressure monitoring for a 24-hr period at the beginning and the end of the 8-week treatment.
4. Patient must be able to communicate and comply with all study requirements and demonstrate good medication compliance.

Exclusion Criteria:

1. Patients with severe hypertension.
2. Patients with history of angioedema, drug-related or otherwise
3. Pregnant or nursing women
4. Women of child-bearing potential , who do not use adequate birth control methods
5. History or evidence of a secondary form of hypertension.
6. History of angina pectoris, myocardial infarction, coronary bypass surgery, ischemic heart disease, surgical or percutaneous arterial intervention of any kind, stroke, TIA, carotid artery stenosis, aortic aneurysm, or peripheral arterial disease.
7. Diabetes mellitus.
8. Previous or current diagnosis of heart failure (NYHA Class II-IV).
9. Clinically significant valvular heart disease at the time of screening.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- China (5):
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
- Japan (10):
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Kunitachi, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- South Korea (5):
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Koyang, Kyunggi
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Seoul
- Taiwan (3):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Changhua
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai

REFERENCES:
- [Derived] Andersen MB, Simonsen U, Wehland M, Pietsch J, Grimm D. LCZ696 (Valsartan/Sacubitril)--A Possible New Treatment for Hypertension and Heart Failure. Basic Clin Pharmacol Toxicol. 2016 Jan;118(1):14-22. doi: 10.1111/bcpt.12453. Epub 2015 Sep 4. PMID 26280447
- [Derived] Kario K, Sun N, Chiang FT, Supasyndh O, Baek SH, Inubushi-Molessa A, Zhang Y, Gotou H, Lefkowitz M, Zhang J. Efficacy and safety of LCZ696, a first-in-class angiotensin receptor neprilysin inhibitor, in Asian patients with hypertension: a randomized, double-blind, placebo-controlled study. Hypertension. 2014 Apr;63(4):698-705. doi: 10.1161/HYPERTENSIONAHA.113.02002. Epub 2014 Jan 20. PMID 24446062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study comprised 3 periods: a 4 week washout and placebo run-in period, an 8 week randomized, double-blind period and a 1 week single-blind, placebo withdrawal period.
Pre-assignment Details: In the run-in period, 457 participants were enrolled. Of the 457 participants, 389 participants were eligible for randomization and randomized in a 1:1:1:1 ratio to each treatment group.
Period: Overall Study
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Started | 100 | 101 | 96 | 92
Full Analysis Set | 100 | 101 | 96 | 92
Placebo Withdrawal Set | 95 | 94 | 93 | 80
Completed | 95 | 94 | 93 | 80
Not Completed | 5 | 7 | 3 | 12
Not completed — Adverse Event | 0 | 1 | 1 | 3
Not completed — Lack of Efficacy | 3 | 1 | 0 | 8
Not completed — Withdrawal by Subject | 2 | 4 | 1 | 1
Not completed — Administrative problems | 0 | 0 | 1 | 0
Not completed — Abnormal test procedure results | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo | Total
Number analyzed (Participants) | 100 | 101 | 96 | 92 | 389
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (10.03) | 52.1 (8.82) | 50.9 (9.81) | 50.9 (10.65) | 51.6 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 27 | 23 | 24 | 114
  Male | 60 | 74 | 73 | 68 | 275

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: Sitting BP measurements were performed at screening through the end of the study at every study visit. A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: Participants from the full analysis set (FAS), who had both baseline and week 8 values, were analyzed. The FAS included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Number analyzed (Participants) | 100 | 98 | 96 | 92
mmHg | -11.53 (0.88) | -10.98 (0.89) | -12.45 (0.90) | -3.69 (0.92)

2. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Description: as for outcome 1
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Number analyzed (Participants) | 100 | 98 | 96 | 92
mmHg | -16.83 (1.25) | -17.54 (1.27) | -20.35 (1.28) | -4.97 (1.30)

3. Secondary Outcome: Change From Baseline in 24 Hour Mean Ambulatory DBP and SBP
Description: Hourly mean ambulatory DBP and SBP post-dosing was calculated for each post-dosing hour over 24 hours by taking the average of the readings taken in the corresponding post-dosing hour at randomization and at week 8. A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Number analyzed (Participants) | 81 | 84 | 82 | 73
mmHg
  maDBP | -8.34 (0.50) | -9.33 (0.49) | -9.69 (0.50) | 0.28 (0.52)
  maSBP | -13.07 (0.65) | -15.18 (0.64) | -15.98 (0.65) | 0.19 (0.68)

4. Secondary Outcome: Change From Baseline in Daytime Mean Ambulatory DBP and SBP
Description: Hourly mean ambulatory DBP and SBP post-dosing was calculated for each post-dosing hour over 24 hours by taking the average of the readings taken in the corresponding post-dosing hour at randomization and at week 8. Daytime mean SBP and DBP were the averages of the hourly means between 6 am and 10 pm. A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Number analyzed (Participants) | 81 | 84 | 82 | 73
mmHg
  maDBP | -8.46 (0.81) | -8.65 (0.80) | -9.77 (0.81) | -0.13 (0.85)
  maSBP | -13.29 (1.08) | -14.62 (1.06) | -16.58 (1.08) | 0.01 (1.13)

5. Secondary Outcome: Change From Baseline in Nighttime Mean Ambulatory DBP and SBP
Description: Hourly mean ambulatory DBP and SBP post-dosing was calculated for each post-dosing hour over 24 hours by taking the average of the readings taken in the corresponding post-dosing hour at randomization and at week 8. Nighttime mean SBP and DBP were the averages of the hourly means between 10 pm and 6 am. A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Number analyzed (Participants) | 81 | 83 | 82 | 73
mmHg
  maDBP | -7.96 (0.81) | -10.36 (0.80) | -9.47 (0.81) | 0.97 (0.85)
  maSBP | -12.27 (1.08) | -16.14 (1.07) | -14.65 (1.08) | 0.61 (1.13)

6. Secondary Outcome: Change From Baseline in Mean Sitting Pulse Pressure
Description: Mean sitting pulse pressure is the difference in msSBP and msDBP (msSBP - msDBP). A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Number analyzed (Participants) | 100 | 98 | 96 | 92
mmHg | -5.11 (0.81) | -6.49 (0.83) | -7.82 (0.83) | -1.09 (0.85)

7. Secondary Outcome: Change From Baseline in Mean Ambulatory Pulse Pressure
Description: Mean ambulatory pulse pressure is the difference in maSBP and maDBP (maSBP - maDBP). A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Number analyzed (Participants) | 81 | 84 | 82 | 73
mmHg | -4.68 (0.30) | -5.84 (0.29) | -6.31 (0.30) | -0.08 (0.31)

8. Secondary Outcome: Number of Participants Who Achieved a Successful Response in msDBP
Description: Successful response in msDBP is defined as msDBP <90 mmHg or a reduction ≥ 10 mmHg from baseline.
Time Frame: 8 weeks
Population: Participants from the full analysis set (FAS), who had week 8 values, were analyzed. The FAS included all randomized participants.
Measure: Number; unit: Participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Number analyzed (Participants) | 100 | 98 | 96 | 92
Participants | 65 | 64 | 67 | 24

9. Secondary Outcome: Number of Participants Who Achieved a Successful Response in msSBP
Description: Successful response in msSBP is defined as msSBP <140 mmHg or a reduction ≥ 20 mmHg from baseline.
Time Frame: 8 weeks
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Number analyzed (Participants) | 100 | 98 | 96 | 92
Participants | 59 | 62 | 66 | 27

10. Secondary Outcome: Number of Participants Who Achieved Successful BP Control
Description: BP control is defined as BP < 140/90 mmHg.
Time Frame: 8 weeks
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Number analyzed (Participants) | 100 | 98 | 96 | 92
Participants | 47 | 48 | 52 | 14

11. Secondary Outcome: Trough to Post-dosing Hour Ratio for Change From Baseline in 24-hour Mean Ambulatory DBP
Description: Trough to post-dosing hour ratio at each post-dosing hour = [trough LSM of LCZ696 - trough LSM of placebo]/[post-dosing hour LSM of LCZ696 - post-dosing hour LSM of placebo]
Time Frame: baseline, 8 weeks
Population: Full Analysis Set (FAS): The FAS included all randomized participants.
Measure: Number; unit: ratio
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg
Number analyzed (Participants) | 100 | 98 | 96
ratio
  Hour 1 | 0.95 | 1.32 | 1.28
  Hour 2 | 0.76 | 1.03 | 0.90
  Hour 3 | 0.64 | 1.35 | 0.91
  Hour 4 | 0.77 | 1.30 | 1.18
  Hour 5 | 0.82 | 1.18 | 1.05
  Hour 6 | 0.73 | 1.04 | 1.21
  Hour 7 | 0.68 | 1.00 | 1.03
  Hour 8 | 0.75 | 0.88 | 0.99
  Hour 9 | 0.80 | 1.07 | 1.01
  Hour 10 | 0.76 | 1.15 | 1.11
  Hour 11 | 0.82 | 1.31 | 1.19
  Hour 12 | 0.56 | 0.92 | 0.89
  Hour 13 | 0.67 | 0.86 | 0.88
  Hour 14 | 0.69 | 0.91 | 0.85
  Hour 15 | 0.57 | 0.69 | 0.74
  Hour 16 | 0.58 | 0.65 | 0.80
  Hour 17 | 0.89 | 0.92 | 1.02
  Hour 18 | 0.86 | 0.92 | 1.07
  Hour 19 | 0.83 | 0.99 | 1.13
  Hour 20 | 0.84 | 1.06 | 1.18
  Hour 21 | 0.76 | 1.02 | 1.02
  Hour 22 | 0.98 | 1.09 | 0.80
  Hour 23 | 1.02 | 0.93 | 0.81
  Hour 24 | 1.00 | 1.00 | 1.00

12. Secondary Outcome: Trough to Post-dosing Hour Ratio for Change From Baseline in 24-hour Mean Ambulatory SBP
Description: as for outcome 11
Time Frame: baseline, 8 weeks
Population: Full Analysis Set (FAS) The FAS included all randomized participants.
Measure: Number; unit: ratio
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg
Number analyzed (Participants) | 100 | 98 | 96
ratio
  Hour 1 | 0.98 | 1.29 | 1.16
  Hour 2 | 1.01 | 1.26 | 1.28
  Hour 3 | 0.97 | 1.35 | 1.13
  Hour 4 | 0.89 | 1.21 | 1.24
  Hour 5 | 0.93 | 1.20 | 1.07
  Hour 6 | 0.87 | 1.20 | 1.33
  Hour 7 | 0.69 | 0.89 | 0.97
  Hour 8 | 0.74 | 0.86 | 1.08
  Hour 9 | 0.74 | 0.90 | 0.99
  Hour 10 | 0.84 | 1.17 | 1.14
  Hour 11 | 0.80 | 1.15 | 1.15
  Hour 12 | 0.69 | 1.01 | 1.08
  Hour 13 | 0.87 | 0.92 | 1.21
  Hour 14 | 0.77 | 0.90 | 1.02
  Hour 15 | 0.67 | 0.79 | 1.01
  Hour 16 | 0.84 | 0.80 | 1.14
  Hour 17 | 1.12 | 1.06 | 1.26
  Hour 18 | 1.04 | 1.05 | 1.46
  Hour 19 | 1.14 | 1.16 | 1.41
  Hour 20 | 1.07 | 1.17 | 1.33
  Hour 21 | 1.06 | 1.12 | 1.39
  Hour 22 | 1.21 | 1.44 | 1.13
  Hour 23 | 1.00 | 1.06 | 1.01
  Hour 24 | 1.00 | 1.00 | 1.00

13. Secondary Outcome: Change From Week 8 to Week 9 in msDBP and msSBP After Single-blind Placebo Withdrawal at Week 8
Description: From week 8 to week 9, participants entered a single-blind placebo withdrawal period to assess the effect of LCZ696 on blood pressure following its discontinuation. Participants, who were randomized to the LCZ696 treatment groups, were discontinued from CLCZ696 at the end of week 8 and all 4 treatment groups received single-blind placebo for 1 week post week 8. A positive change from week 8 to week 9 indicates worsening.
Time Frame: 8 weeks, 9 weeks
Population: Only participants from the full analysis, who had values at both week 8 and week 9, were included in the analysis. The FAS included all randomized participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Number analyzed (Participants) | 95 | 94 | 93 | 80
mmHg
  msDBP | 4.8 (7.61) | 5.1 (7.03) | 5.6 (7.01) | -0.6 (6.34)
  msSBP | 8.0 (11.88) | 8.8 (11.62) | 11.6 (10.96) | -0.7 (10.50)

ADVERSE EVENTS:
Arm/Group | LCZ696 100 mg | LCZ696 200 mg | LCZ696 400 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/101 | 2/96 | 0/92
Other Adverse Events (participants affected / at risk) | 16/100 | 11/101 | 14/96 | 15/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 100 mg (N=100) | LCZ696 200 mg (N=101) | LCZ696 400 mg (N=96) | Placebo (N=92)
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 100 mg (N=100) | LCZ696 200 mg (N=101) | LCZ696 400 mg (N=96) | Placebo (N=92)
Nasopharyngitis (Infections and infestations) | 6 | 6 | 7 | 7
Upper respiratory tract infection (Infections and infestations) | 9 | 3 | 4 | 4
Dizziness (Nervous system disorders) | 1 | 2 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.